CLINICAL TRIAL: NCT04066634
Title: Assessment of the Vivio System as an Aid in the Identification of Heart Sounds Associated With Severe Aortic Stenosis
Brief Title: Vivio AS (Aortic Stenosis) Detection Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avicena LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VS-001-AS
Record Dates: First submitted 2019-07-25; First posted 2019-08-26 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Assist in Diagnosis (Experimental): The Vivio Analysis Software is an analysis software that assists in identifying suspected systolic murmurs associated with aortic stenosis. The Vivio Analysis Software is used with the Vivio System, a non-invasive device used for the detection and amplification of sounds from the heart and arteries.
  Interventions: Device: Vivio System

INTERVENTIONS:
Device: Vivio System — The Vivio Analysis Software is an analysis software that assists in identifying suspected systolic murmurs associated with aortic stenosis. The Vivio Analysis Software is used with the Vivio System, a non-invasive device used for the detection and amplification of sounds from the heart and arteries.
  Other Names: Electronic stethoscope

SUMMARY:
Evaluate the sensitivity and specificity of the Vivio System when used as an aid in the identification of heart sounds associated with severe aortic stenosis.

DETAILED DESCRIPTION:
Prospective, non-randomized, multi-center study of adult subjects referred for echocardiography. Total of 200 enrolled subjects at 3 sites. Up to 10 roll-in subjects per site. Enrolled subjects will undergo: Vivio data capture, Eko stethoscope capture of heart sounds, Standard of care transthoracic echocardiogram (TTE). Vivio analysis will not be available to non-Avicena personnel. Recorded sounds from the FDA-approved Eko stethoscope will be presented to an independent expert physician review panel blinded to Vivio and TTE results, to compare diagnosis of severe AS using Eko (auscultation) vs. Vivio (algorithms).

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (21 years of age or older).
2. Referred for transthoracic echocardiography by physician/primary care provider/cardiologist.
3. Willing and able to participate in all study evaluations and allow access to medical testing and records.
4. Signed informed consent or have a legally authorized representative who provides informed consent on behalf of the subject.

Exclusion Criteria:

1. Acute coronary syndrome, cardiogenic shock or the need for inotropic/mechanical circulatory support.
2. Need for bedside echocardiogram (inpatient).
3. Prosthetic device previously implanted at aortic valve position.
4. Inability to palpate carotid pulse (e.g. due to severe obesity)
5. History of carotid sinus hypersensitivity (i.e. fainting in response to touching or positioning the neck).
6. History of carotid artery disease or treatment (e.g. unstable carotid plaques that might rupture upon massage or endarterectomy).
7. Open skin lesions at target site of electronic stethoscope/Vivio device examination.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint - Sensitivity and specificity of detection of heart sounds associated with severe aortic stenosis by the Vivio System | 48 Hours
  Sensitivity and specificity of detection of heart sounds associated with severe aortic stenosis by the Vivio System compared to the Expert Physician Panel (EPP).

SECONDARY OUTCOMES:
Secondary Endpoint 1 - Sensitivity and specificity relative to PCPP detection of heart sounds associated with severe aortic stenosis. | 48 Hours
  Sensitivity and specificity relative to PCPP detection of heart sounds associated with severe aortic stenosis.
Secondary Endpoint 2 - Correlation of Vivio results to transthoracic echocardiography assessment of aortic stenosis as determined by echocardiography. | 48 Hours
  Correlation of Vivio results to transthoracic echocardiography assessment of aortic stenosis as determined by echocardiography.
Secondary Endpoint 3 - Additional analysis of data to include Likelihood Ratios (LR), Positive Predictive Value (PPV), and Negative Predictive Value (NPV). | 48 Hours
  Additional analysis of data to include Likelihood Ratios (LR), Positive Predictive Value (PPV), and Negative Predictive Value (NPV).
Secondary Endpoint 4 - Assessment of type and degree of all heart sounds associated with aortic stenosis (mild/moderate/severe). | 48 Hours
  Assessment of type and degree of all heart sounds associated with aortic stenosis (mild/moderate/severe). The heart sounds associated with severe aortic stenosis using a traditional electronic stethoscope include S1 (normal), S2 (single or paradoxically split) and a late peaking (mid to late systole) diamond shaped, grade 3 or higher murmur. The Vivio system can detect a single component of S2 (aortic) over the carotid but not the pulmonic component or splitting characteristics. It can also detect the nature and timing of the systolic murmur as transmitted through the vascular system to the carotid. The heart sounds associated with severe aortic stenosis include S1 (normal), presence or absence of S2. Less severe aortic stenosis is characterized by an early to mid-peaking diamond shape murmur with a soft but present aortic component of S2.

OTHER OUTCOMES:
Ancillary Endpoint - Incidence of Adverse Events | 48 Hours
  Incidence of Adverse Events: Summary of all reported adverse events during the study. Events will be summarized by seriousness (e.g. serious vs. non-serious), attribution (e.g. device vs. procedure vs. comorbidity) based upon site reported data.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Brady, JD, Study Director — Avicena LLC
Locations (3):
- United States (3):
  - Morristown Medical Center, Morristown, New Jersey
  - St. Francis Hospital, Roslyn, New York
  - Miriam Hospital, Providence, Rhode Island